CLINICAL TRIAL: NCT00765570
Title: Treatment of Advanced Bulky Malignancies With Spatially Fractioned Radiation Therapy A Phase II Randomized Trial
Brief Title: Study of Advanced Bulky Malignancies With Spatially Fractioned Radiation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual too slow - would not enroll enough subjects to determine outcome
Sponsor: Summa Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRID
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-04

CONDITIONS: Advanced Bulky Malignancies
Keywords: large tumors in the head & neck, lung, abdomen or pelvis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Active Comparator): Treatment Group 1-one treatment of Grid therapy followed by 15 treatments with standard radiation
  Interventions: Radiation: Spatially Fractioned Radiation Therapy; Radiation: Treatment Group 1
- Treatment Group-2 (Active Comparator): Treatment Group 2-15 treatments with standard radiation
  Interventions: Radiation: Standard radiation

INTERVENTIONS:
Radiation: Spatially Fractioned Radiation Therapy — evaluate response to radiation therapy by a large bulky tumor influenced by adding a single dose of 15 Gy grid radiotherapy.
  Other Names: GRID Radiation
  Arms: Treatment Group 1
Radiation: Treatment Group 1 — one treatment of Grid therapy followed by 15 treatments with standard radiation
  Arms: Treatment Group 1
Radiation: Standard radiation — 15 Standard radiation treatments
  Other Names: Treatment Group 2
  Arms: Treatment Group-2
Radiation: Standard radiation — standard radiation treatment
  Other Names: Treatment Group 2
  Arms: Treatment Group-2

SUMMARY:
Expand clinical literature on the use of Grid radiation with conventional external beam therapy. Vast majority of therapy is for palliative care to provide relief from pain, but has also shown a reduction in the size of tumor mass.

DETAILED DESCRIPTION:
This study will evaluate response to radiation therapy by a large bulky tumor is influenced by adding a single dose of 15 Gy grid radiotherapy. To accomplish this, patients with large bulky tumors in the lung, abdomen or pelvis will be randomized to receive either standard palliative radiation or palliative radiation plus a single fraction of grid radiation. Tumor response, pain relief and duration of response, and pain control will be monitored. Toxicity of treatment will also be followed. The hypothesis of this study is that grid radiation will produce a significant improvement in tumor response and pain control that produces no further increase in acute or late toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic or cytologic diagnosis of primary or metastatic epithelial cancer or sarcoma located in the head and neck area, lung, abdomen or pelvis.
* Tumors must have an overall dimension greater than 24 cm2 (bidimensional) with one dimensions >6 cm, by x-ray, CT/MRI scan or clinical exam.
* Age >18
* Karnofsky > 70 with life expectancy >3 months.
* Patients may not begin new hormone therapy within 2 weeks of initiation of protocol treatment.
* No planned initiation of hormone therapy within 2 weeks of protocol therapy
* Adequate bone marrow function: Hb > 9, white blood cell count (WBC) > 2,000. Hepatic function < 3x upper limit of laboratory normal values.
* Laboratory studies will be obtained within 2 weeks prior to randomization.
* Patients with metastatic sites of disease including brain are eligible provided that life expectancy is > 3 months.

Exclusion Criteria:

* Hematologic-related tumors.
* Tumors overlying critical central nervous system structures including spinal cord, eye or brainstem or require treatment portals over these vital structures.
* Central nervous system tumors
* Evidence of other primary malignancy except for carcinoma in situ of cervix or skin cancer excluding melanoma unless disease free for 2 years prior to randomization
* Patients with spinal cord compression.
* Prior radiation to treatment field.
* Concomitant chemotherapy or chemotherapy within past 2 weeks. Planned initiation of chemotherapy within 2 weeks of completing protocol treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seider, Ph.D., M.D., Principal Investigator — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled from the physicians offices at Summa Health System.
Groups:
- Treatment Group-2: Treatment Group 2:15 treatments with standard radiation
Period: Overall Study
Arm/Group | Treatment Group 1 | Treatment Group-2
Started | 9 | 3
Completed | 7 | 3
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group-2: Treatment Group 2: 15 treatments with standard radiation
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 | Treatment Group-2 | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (12) | 69 (9) | 72 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Protocol Treatment Related Morbidity
Description: Number of grade 3 or higher complications during the assesment period. This does not include any complication felt to be due solely to malignancy
Time Frame: during duration of treatment of 3 weeks. Follow up exams every 6 months for the next two years and then yearly for the rest of your life.
Measure: Number; unit: events
Arm/Group | Treatment Group 1 | Treatment Group-2
Number analyzed (Participants) | 9 | 3
events
  Grade 3 Adverse Events | 0 | 0
  Grade 4 Adverse Events | 0 | 0
  Grade 5 Adverse Events | 0 | 0

2. Secondary Outcome: Objective Response of Bulky Tumors of the Head and Neck Area, Lung, Abdomen or Pelvis to Standard Fractionated Radiation Therapy Plus Grid Therapy Compared to Standard Fractionated Radiation Therapy Alone.
Description: Complete response (CR) = 100% tumor disappearance Partial response (PR) = > 50% reduction in size Stable disease (SD) = < 50% reduction or no change +/- 10% increase in tumor size Progressive disease (PD) = > 10% increase in size of tumor Unknown Status (UK)
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Treatment Group 1 | Treatment Group-2
Number analyzed (Participants) | 9 | 3
participants
  Complete Response (CR) | 1 | 0
  Partial response (PR) | 0 | 1
  Stable disease (SD) | 6 | 2
  Progressive disease (PD) | 1 | 0
  Unknown (UK) | 1 | 0

ADVERSE EVENTS:
Time Frame: Patients were to be assessed at 2 weeks, 4 weeks, 8 weeks, 12 weeks, 6 months, 9 months and 1 year after treatment was completed. Follow-up after 1 year was to be at 6 month intervals until 2 years, then annually.
Arm/Group | Treatment Group 1 | Treatment Group-2
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 8/9 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 (N=9) | Treatment Group-2 (N=3)
Skin Toxicity (Skin and subcutaneous tissue disorders) | 6 | 2
Lung Toxicity (Respiratory, thoracic and mediastinal disorders) | 4 | 1 — cough, dyspnea
CNS Toxicity (Nervous system disorders) | 1 | 0
GI or GU Toxicity (Gastrointestinal disorders) | 3 | 0
other (General disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No